CLINICAL TRIAL: NCT06424990
Title: Biodex Balance Training With Transcutaneous Electrical Nerve Stimulation for Children With Spastic Diplegia: A Double-blinded, Randomized, Placebo-controlled Trial
Brief Title: Balance Training With TENS for Spastic Diplegic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: balancing with TENS for CP
Record Dates: First submitted 2024-05-11; First posted 2024-05-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: balance training with TENS
- control group (Placebo Comparator)
  Interventions: Other: Balance training with placebo TENS

INTERVENTIONS:
Other: balance training with TENS — children will receive Biodex balance training with TENS for 30 minutes a day, 5 days per week for 4 weeks
  Arms: study group
Other: Balance training with placebo TENS — children will receive Biodex balance training with placebo TENS for the same period.
  Arms: control group

SUMMARY:
Children with spastic diplegic Cerebral Palsy (CP) often show motor impairment due to a number of deficits; including poor muscle control, weakness, spasticity and reduced range of motion in the extremities. All these factors affect the ability of children with CP to maintain balance and walk which are the primary rehabilitation concerns of parents and clinicians. The Balance Trainer provides a safe balance environment and assists with muscle activation of ankle and hip joints, and it is hypothesized that to promote spasticity inhibition, the use of TENS may decrease hyper-excitability, modulate reciprocal inhibition, and increase presynaptic inhibition. To the best of the authors' knowledge, the current study is the first research to investigate the effect of using Biodex balance training with TENS in improving children with spastic diplegia.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of spastic diplegia cerebral palsy.
* Age from 10 to 12 years.
* Spasticity grade 1 and 1+ according to the Modified Ashworth scale.
* Level II motor function according to the Growth Motor Function Classification System.
* Able to understand and follow instructions.
* Their heights are more than 100 cm and weights are more than 20 Kg which are the lower limits of height and weight needed by the Biodex stability system.

Exclusion Criteria:

* Epilepsy.
* Significant visual or auditory problems according to medical reports (audio-vestibular and ophthalmic examination).
* Structural or fixed soft tissue deformities of the lower extremities.
* Neurological or orthopedic surgery in the past 12 months.
* Botox injection in the lower extremities in the past 6 months.
* Fracture, sprain, or strain injury of the lower extremities in the past 6 months.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
hip adductor spasticity | change from base line at 4 weeks.
  spasticity of hip adductors will be measured by the Modified Ashworth Scale. Modified ashworth scale grades of spasticity are as follows: 0 = normal muscle tone; 1= slight increase in muscle tone, manifested by catch and release or by minimal resistance at the end; 1+ = slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout; 2= more marked increase in muscle tone, but limb easily flexed; 3= considerable increase in muscle tone, passive movement difficult; and 4 = limb rigid in flexion or extension.
spatio-temporal gait parameters | change from base line at 4 weeks.
  Spatiotemporal gait parameters (Walking Speed (WS) (m/s), Step Length (SL) (cm) and the Stance Time (ST) (%) on each limb) using GAITRite system which has excellent reliability for measuring most spatio-temporal gait parameters. The GAITRite is a 700 cm × 90 cm electronic walkway with an active sensor area of 610 cm long and 60 cm wide. The active area contains 23,040 embedded pressure-activated sensors with a spatial resolution of 1.27 cm and a sampling rate of 120 Hz. All data was processed and stored by an IBM compatible computer using GAITRite® gold, Version 3.2b software.
balance assessment | change from base line at 4 weeks
  anteroposterior stability index, mediolateral stability index, and overall stability index will be measured using Biodex balance system. Biodex Stability System has an intertester intraclass correlation coefficients (ICCs) equals 0.70 and an intratester ICCs equals 0.82. Biodex Stability System formed of a dynamic platform that allows movements to occur around the anterior-posterior (AP) and mediallateral (ML) axes simultaneously. Biodex Stability System has a screen displaying the child's position on it and a support handle that can be adjusted according to each child's height. The screen gives visual feedback about the degree of tilting that helps the child to maintain the cursor in the center of the screen to obtain a good score of balance. The higher the scores, the poorer the balance of the child

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt